CLINICAL TRIAL: NCT04108858
Title: Phase Ib/II Trial of Copanlisib in Combination With Trastuzumab and Pertuzumab After Induction Treatment of HER2 Positive (HER2+) Metastatic Breast Cancer (MBC) With PIK3CA Mutation or PTEN Mutation
Brief Title: Testing the Addition of an Anti-cancer Drug, Copanlisib, to the Usual Maintenance Treatment (Trastuzumab and Pertuzumab) After Initial Chemotherapy in a Phase Ib/II Trial for Advanced HER2 Positive Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-06461; NCI-2019-06461 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MDACC# 2020-0260; 10296 (Other: University of Texas MD Anderson Cancer Center LAO); 10296 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; HER2-Positive Breast Carcinoma; Metastatic Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — copanlisib; pertuzumab; 2C4 antibody; Trastuzumab; CT-P6; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I, Phase II Arm I (copanlisib, trastuzumab, pertuzumab) (Experimental): Patients receive copanlisib IV over 60 minutes on days 1 and 8. Patients also receive trastuzumab IV over 30-90 minutes and pertuzumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Copanlisib; Biological: Pertuzumab; Biological: Trastuzumab
- Phase II Arm II (trastuzumab, pertuzumab) (Active Comparator): Patients receive trastuzumab IV over 30-90 minutes and pertuzumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pertuzumab; Biological: Trastuzumab

INTERVENTIONS:
Drug: Copanlisib — Given IV
  Other Names: BAY 80-6946; PI3K Inhibitor BAY 80-6946
  Arms: Phase I, Phase II Arm I (copanlisib, trastuzumab, pertuzumab)
Biological: Pertuzumab — Given IV
  Other Names: 2C4; 2C4 Antibody; BCD-178; EG1206A; HLX11; HS627; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; Pertuzumab Biosimilar BCD-178; Pertuzumab Biosimilar EG1206A; Pertuzumab Biosimilar HLX11; Pertuzumab Biosimilar HS627; Pertuzumab Biosimilar TQB2440; Rhumab 2C4; rhuMAb2C4; RO4368451; TQB 2440; TQB-2440; TQB2440
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Biceltis; CANMab; CT-P06; CT-P6; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herclon; Hertraz; Herzuma; Kanjinti; Ogivri; Ontruzant; PF-05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; Trastuzumab Biosimilar CT-P6; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of copanlisib when given together with trastuzumab and pertuzumab and to see how well they work after induction treatment in treating patients with HER2 positive stage IV breast cancer with PIK3CA or PTEN mutation. Copanlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Trastuzumab is a form of "targeted therapy" because it works by attaching itself to specific molecules (receptors) on the surface of cancer cells, known as HER2 receptors. When trastuzumab attaches to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by the body's immune system. Monoclonal antibodies, such as pertuzumab, may kill tumor cells that are left after chemotherapy. The addition of copanlisib to the usual treatment (trastuzumab and pertuzumab) could shrink the cancer or stabilize it for longer duration as compared to the usual treatment alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and recommended phase 2 dose (RP2D) of the combination of copanlisib, trastuzumab and pertuzumab in patients with metastatic epidermal growth factor receptor 2 (HER2)-positive breast cancer. (Phase Ib) II. To assess the benefit of adding copanlisib to trastuzumab and pertuzumab in HER2-positive metastatic breast cancer patients with PIK3CA mutations or PTEN mutation receiving maintenance therapy after induction treatment, as measured by progression free survival (PFS). (Phase II)

SECONDARY OBJECTIVES:

I. To assess the benefit of adding copanlisib to trastuzumab and pertuzumab in HER2-positive metastatic breast cancer patients with PIK3CA mutations or PTEN mutation receiving maintenance therapy after induction treatment, as measured by overall survival (OS). (Phase II) II. To evaluate the safety of copanlisib given at the RP2D in combination with trastuzumab and pertuzumab. (Phase II)

EXPLORATORY OBJECTIVES:

I. To correlate PFS and OS of the patients who receive the triplet combination with:

Ia. The number of induction cycles. Ib. Hormone receptor status (estrogen receptor [ER] and progesterone receptor [PR]).

Ic. PTEN loss by immunohistochemistry (IHC). Id. PIK3CA mutations or PTEN mutations. (Phase Ib)

II. To assess PTEN IHC, Ki-67 IHC and cleaved caspase-3 IHC and to perform molecular profiling assays on malignant and normal tissues, including, but not limited to, whole exome sequencing (WES) and messenger ribonucleic acid (RNA) sequencing (RNAseq), in order to:

IIa. Identify potential predictive and prognostic biomarkers associated with treatment outcomes (PFS and OS) with the addition of copanlisib to dual HER2-targeted treatment.

IIb. Identify resistance mechanisms using genomic deoxyribonucleic acid (DNA)- and RNA-based assessment platforms.

III. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

IV. To bank formalin-fixed, paraffin-embedded (FFPE) tissue, blood (for cell-free DNA analysis), and nucleic acids obtained from patients at the Experimental Therapeutics Clinical Trials Network (ETCTN) Biorepository at Nationwide Children's Hospital.

OUTLINE:

PHASE I: Patients receive copanlisib intravenously (IV) over 60 minutes on days 1 and 8. Patients also receive trastuzumab IV over 30-90 minutes and pertuzumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive copanlisib IV over 60 minutes on days 1 and 8. Patients also receive trastuzumab IV over 30-90 minutes and pertuzumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive trastuzumab IV over 30-90 minutes and pertuzumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1B: Any prior number of lines of therapy in metastatic setting is allowed, provided patients are considered candidates for trastuzumab and pertuzumab combination or on maintenance trastuzumab and pertuzumab (with or without prior chemotherapy) as long as dose limiting toxicity (DLT) can be determined. For Phase 2:Patients should have only received first line of induction chemotherapy (taxane) with trastuzumab and pertuzumab in the metastatic setting
* Presence of actionable mutation in either PIK3CA or PTEN on molecular testing
* For Phase 2-Patients must be within 8 weeks of completion of first-line induction chemotherapy (i.e., 4-8 cycles of any taxane, trastuzumab and pertuzumab) without evidence of progression. Patients may receive up to 2 doses of HER2 targeted treatment between end of induction treatment and start of trial, while eligibility is being confirmed
* Clinical stage IV as assessed by American Joint Committee on Cancer (AJCC) (8th edition, anatomic staging) guidelines with known metastatic disease (Edge and Compton, 2010; Amin et al., 2017)
* HER2+ breast cancer patients with any ER/PR status as assessed by the American Society of Clinical Oncology (ASCO)-College of American Pathologists (ASCO-CAP) guidelines (Wolff et al., 2013; Wolff et al., 2018). HER2 testing of metastasis will be required
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Left ventricular ejection fraction (LVEF) >= 50% by echocardiogram or multigated acquisition scan (MUGA)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN OR =< 5 x ULN for subjects with liver metastases
* Creatinine =< 1.5 x institutional ULN OR measured or calculated creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]). Creatinine clearance should be calculated per institutional standard
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless patient is receiving anticoagulation as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless patient is receiving anticoagulation as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Patients with treated brain metastases are eligible if follow-up brain imaging 30 days after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients who are therapeutically treated with anticoagulation including warfarin will be allowed to participate provided that their medication dose and INR/PTT is stable. Due to interaction of copanlisib with warfarin, patients who are on warfarin should be monitored closely while on this trial
* Women of child-bearing potential MUST have a negative serum or urine human chorionic gonadotropin (HCG) test unless prior tubal ligation (>= 1 year before screening), total hysterectomy or menopause (defined as 12 consecutive months of amenorrhea). Patients should not become pregnant or breastfeed while on this study
* Patients and their partners, if sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for 7 months after last dose of study drug(s) to prevent pregnancy in the study patient or partner
* Hormone receptor positive (ER+ and / PR+) breast cancer patients will be allowed to continue endocrine therapy as clinically indicated while participating in the study.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Known active hepatitis B or hepatitis C infection. All patients must be screened for hepatitis B virus (HBV) and hepatitis C virus (HCV) up to 28 days prior to study drug start using the routine hepatitis virus lab panel. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on non-CYP3A4-interactive suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV ribonucleic acid (RNA)
* Human immunodeficiency virus (HIV)-positive patients, unless they have CD4 counts > 500 cells/mm^3 in the past 6 months and do not require CYP3A4-interactive antiretroviral therapy
* Active infection requiring IV antibiotics or other uncontrolled intercurrent illness requiring hospitalization
* Inability to comply with the study and follow-up procedures
* History of cerebrovascular accident (CVA), myocardial infarction, symptomatic congestive heart failure, cardiac arrhythmia, or unstable angina within the previous 6 months before starting therapy
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the following exceptions: alopecia (any grade is acceptable); neuropathy must have resolved to =< grade 2. Congestive heart failure (CHF) due to prior anti-cancer therapy must have been =< grade 1 in severity at the time of occurrence, and must have resolved completely
* Current uncontrolled hypertension (>= 150/90)
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has a known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Patients with uncontrolled type I or II diabetes mellitus (DM); uncontrolled DM is defined as glycosylated hemoglobin (HbA1c) > 8.5% and a fasting blood glucose of > 120 mg/dL within 14 days prior to trial entry
* Immunosuppressive therapy is not allowed while on study
* Patients who are receiving any other investigational agents
* Patients with leptomeningeal disease or active untreated brain metastases
* Prior exposure to any PI3K, AKT or mTOR inhibitors. History of allergic reactions attributed to compounds of similar chemical or biologic composition to copanlisib, PI3K inhibitors, or HER2 inhibitors
* Copanlisib is primarily metabolized by CYP3A4. Therefore, the concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and strong inducers of CYP3A4 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's wort) are not permitted from 14 days prior to enrollment until the end of the study. Other medications that are prohibited while on copanlisib treatment:

  * Herbal medications/preparations (except for vitamins)
  * Anti-arrhythmic therapy other than beta blockers or digoxin
  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Systemic corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not permitted while on study. Previous corticosteroid therapy must be stopped or reduced to the allowed dose at least 7 days prior to the computed tomography (CT)/magnetic resonance imaging (MRI) screening. If a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose before the screening. Patients may be using topical or inhaled corticosteroids
* Patients with non-healing wound, ulcer, or bone fracture
* Pregnant women are excluded from this study because copanlisib is a PI3K inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with copanlisib, breastfeeding should be discontinued if the mother is treated with copanlisib. These potential risks may also apply to other agents used in this study
* Patients are eligible to receive standard of care therapy that would confer clinical benefit to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Damodaran, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (5):
- United States (5):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Any participants referred was screened for eligibility. Participants with required mutation were the only participants referred.
Pre-assignment Details: No exclusions to report.
Groups:
- Phase 1, Dose Level 1: Copanlisib 60mg given D1 and D8 over 60mins of each cycle+ trastuzumab, pertuzumab given over 30mins D1 of each cycle all drugs given IV infusion each cycle is 21 days
Period: Overall Study
Arm/Group | Phase 1, Dose Level 1
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: This clinical trial did not attract participants who met the eligibility criteria, resulting in poor accrual.
Arm/Group | Phase 1, Dose Level 1
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety run-in Phase 1b/2
Description: Incidence of adverse events and serious adverse events to determine safety: incidence of DLTs to determine RP2D
Time Frame: 21 days
Population: This clinical trial did not attract participants who met the eligibility criteria, resulting in poor accrual. Stopped during Phase 1 portion and did not proceed to Phase 2.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Arm II (Copanlisib, Trastuzumab, Pertuzumab): Participants receive copanlisib IV over 60 minutes on days 1 and 8. Participants also receive trastuzumab IV over 30-90 minutes and pertuzumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Copanlisib: Given IV Pertuzumab: Given IV Trastuzumab: Given IV
Arm/Group | Phase 1, Dose Level 1 | Phase II Arm II (Copanlisib, Trastuzumab, Pertuzumab)
Number analyzed (Participants) | 2 | 0
Participants | 2 |

2. Primary Outcome: Incidence of Dose Limiting Toxicities (DLTs) (Phase Ib)
Time Frame: 21 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Phase Ib/II Trial of Copanlisib in Combination With Trastuzumab and Pertuzumab in HER2 Positive MBC: Participants receive copanlisib IV over 60 minutes on days 1 and 8. Participants also receive trastuzumab IV over 30-90 minutes and pertuzumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Copanlisib: Given IV
  Pertuzumab: Given IV
  Trastuzumab: Given IV
Arm/Group | Phase Ib/II Trial of Copanlisib in Combination With Trastuzumab and Pertuzumab in HER2 Positive MBC
Number analyzed (Participants) | 2
Participants | 0

3. Primary Outcome: Progression-free Survival (PFS) (Phase II)
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Phase Ib/II Trial of Copanlisib in Combination With Trastuzumab and Pertuzumab in HER2 Positive MBC | Phase II Arm II (Copanlisib, Trastuzumab, Pertuzumab)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression-free Survival (Phase Ib)
Time Frame: 12 months
Population: This clinical trial did not attract participants who met the eligibility criteria, resulting in poor accrual. Stopped during Phase 1 portion and did not proceed to Phase 2. We had a total of two participants enrolled in the escalation phase. Patient 1 was on study for 9 weeks and patient 2 was on study for 18 weeks. Study was closed due to poor accrual. No data for analysis.
Arm/Group | Phase Ib/II Trial of Copanlisib in Combination With Trastuzumab and Pertuzumab in HER2 Positive MBC | Phase II Arm II (Copanlisib, Trastuzumab, Pertuzumab)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS) (Phase Ib)
Time Frame: 12 months
Population: This clinical trial did not attract participants who met the eligibility criteria, resulting in poor accrual. Stopped during Phase 1 portion and did not proceed to Phase 2. We had a total of two participants enrolled in the escalation phase. Since study was prematurely terminated due to poor accrual formal OS analysis could not be performed. No data for analysis.
Arm/Group | Phase Ib/II Trial of Copanlisib in Combination With Trastuzumab and Pertuzumab in HER2 Positive MBC | Phase II Arm II (Copanlisib, Trastuzumab, Pertuzumab)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Survival (OS) (Phase II)
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Phase Ib/II Trial of Copanlisib in Combination With Trastuzumab and Pertuzumab in HER2 Positive MBC | Phase II Arm II (Copanlisib, Trastuzumab, Pertuzumab)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Adverse Events and Serious Adverse Events (Phase II)
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Phase Ib/II Trial of Copanlisib in Combination With Trastuzumab and Pertuzumab in HER2 Positive MBC | Phase II Arm II (Copanlisib, Trastuzumab, Pertuzumab)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 months
Description: This clinical trial did not attract participants who met the eligibility criteria, resulting in poor accrual.
Groups:
- Phase 1, Dose Level 1: Copanlisib 60 mg given D1 and D8 of each 21 day cycle +Trastuzumab, pertuzumab given D1 of each 21 day cycle
Arm/Group | Phase 1, Dose Level 1
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1, Dose Level 1 (N=2)
Diarrhea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
aPTT (Investigations) | 1
Alk phos (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Blurred vision (Eye disorders) | 1
bruising (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Dyspena (Respiratory, thoracic and mediastinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
oral mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Papulopustular (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT04108858/Prot_SAP_000.pdf
  • Informed Consent Form: Phase I Informed Consent Form (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT04108858/ICF_001.pdf
  • Informed Consent Form: Phase II Informed Consent Form (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT04108858/ICF_002.pdf